CLINICAL TRIAL: NCT00002081
Title: Open-Label Program of Dideoxycytidine ( ddC ) to Be Used in Combination With Zidovudine ( AZT ) for Treatment of Advanced HIV Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 031E; NV14147C
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1992-06

CONDITIONS: HIV Infections
Keywords: Zalcitabine; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Zidovudine; Zalcitabine

INTERVENTIONS:
Drug: Zidovudine
Drug: Zalcitabine

SUMMARY:
To provide zalcitabine ( dideoxycytidine; ddC ) for use with zidovudine ( AZT ) in patients with advanced HIV infection. To observe serious toxicities in this population.

DETAILED DESCRIPTION:
Patients are treated with 1 of 2 doses of ddC administered orally (PO) in combination with AZT administered PO (patients who are unable to tolerate this dose of AZT may receive a lower dose).

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Concomitant use of investigational compounds for prophylaxis or treatment of opportunistic infections or other treatments provided use of those compounds with ddC-AZT is considered safe.

Patients must have:

* Documented HIV infection OR documented AIDS-defining opportunistic infection or neoplasm.
* Previous AIDS-defining opportunistic infection, neoplasm, or condition OR CD4 lymphocyte count equal to or less than 300 cells/mm3 if symptomatic ORCD4 lymphocyte count equal to or less than 200 cells/mm3 if asymptomatic.
* Patients must not be currently enrolled in or must be unable to enter an AIDS Clinical Trials Group (ACTG), Community Programs for Clinical Research on AIDS (CPCRA), or other controlled clinical program because of patient ineligibility, distance from trial site, or patient refusal.
* Patients currently enrolled in any controlled clinical trial of an anti-HIV compound may enter this program only if they have met the end points required for termination of that trial.
* Patients may be co-enrolled in clinical programs of investigational compounds being tested for prophylaxis or treatment of opportunistic infections or other treatments provided that program allows ddC-AZT combination use, and concomitant administration of the other investigational drug and ddC-AZT is considered safe by the investigator.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Any clinical or laboratory toxicity or abnormality, particularly the presence or history of moderate to severe peripheral neuropathy, that would pose an undue risk to the patient upon initiation of ddC-AZT treatment.
* Pregnancy.

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- ddC Coordinating Ctr, Wellesley Hills, Massachusetts, United States

REFERENCES:
- [Background] Walker M, Moyle GJ, Harris R, Warburg M. Safety and efficacy of zalcitabine (ddC) and zidovudine (ZDV) combination in HIV-positive persons with CD4 cell counts less than or equal to 300/mm3: an international open label evaluation (Roche study M50002). Int Conf AIDS. 1996 Jul 7-12;11(1):77 (abstract no MoB1129)